CLINICAL TRIAL: NCT02714205
Title: Flushing Reduction Associated With Nitrates
Acronym: FRAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alison Huang, MD (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Alison Huang, MD, Associate Professor of Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-18472; 5R01AG050588-04 (NIH)
Record Dates: First submitted 2016-03-11; First posted 2016-03-21 (Estimated); Results first posted 2023-05-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Menopausal Hot Flashes
Keywords: Hot flash
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Transdermal Nitroglycerin (Experimental): Daily transdermal nitroglycerin patch, starting at 0.2 mg/hr. Dose escalation up to 0.6 mg/hr.
  Interventions: Drug: transdermal nitroglycerin
- Placebo (Placebo Comparator): Daily transdermal placebo patch.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: transdermal nitroglycerin — Study participants will be randomized to transdermal nitroglycerin patch or placebo patch. Participants will wear a study medication patch daily, for 12 weeks.
  Arms: Transdermal Nitroglycerin
Drug: Placebo — Study participants will be randomized to transdermal nitroglycerin patch or placebo patch. Participants will wear a study medication patch daily, for 12 weeks.
  Arms: Placebo

SUMMARY:
A randomized, double-blinded, placebo-controlled trial of uninterrupted transdermal nitrate therapy in 140 peri- or postmenopausal women who have frequent hot flashes. Women will be randomly assigned to uninterrupted use of transdermal nitrate therapy (participant directed dose-escalation of 0.2 to 0.6 mg/hr) or identical-appearing placebo patches for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40 to 62 years (consistent with the recent MSFlash hot flash network trials, and likely to maximize enrollment of highly symptomatic women)
* Postmenopausal or in the late menopausal transition. For this study, postmenopausal status will be defined by: 1) self-reported history of bilateral oophorectomy, 2) follicle stimulating hormone (FSH) levels > 20 mU/mL for those with a self-reported history of hysterectomy without bilateral oophorectomy, or 3) no self-reported history of hysterectomy or oophorectomy, but absence of menses in the past 12 months. Late menopausal transition will be defined by amenorrhea for at least 60 days in the past 12 months within the specified age group.
* Documentation of an average of 7 or more hot flashes per 24 hours as well as 4 or more moderate-to-severe hot flashes per 24 hours as recorded on a validated 7-day screening symptom diary
* Willing to refrain from initiating other treatments that are known to affect the frequency of severity hot flashes during the trial period
* Report having a current primary health care provider (such as a general practitioner, family medicine, internal medicine, or nurse practitioner providing primary care or specializing in women's health)

Exclusion Criteria:

* Current or recent use of NTG or other nitrate-containing medications (i.e., use within 1 month of screening), or intention to use nitrate-containing medication during the interventional period
* Current or recent use of medications already known to reduce the frequency or severity of hot flashes (e.g., vaginal or transdermal estrogens in the past 4 weeks; oral estrogens or progestins in the past 8 weeks; intrauterine progestin therapy in the past 8 weeks; progestin implants or estrogen alone injectable therapy in the past 3 months; estrogen pellet therapy or progestin injectable therapy in the past 6 months; clonidine, methyldopa, gabapentin, pregabalin and selective serotonin or norepinephrine reuptake inhibitors (SSRIs/SNRIs) in the past 1 month); or intention to use these medications during the interventional period
* Current or recent use of phosphodiesterase inhibitor medications (within 1 month of screening), or intention to use these medications during the interventional period
* Current or recent use of riociguat, a soluble guanylate cyclase stimulator medication, within 1 month of screening, or intention to use riociguat during the interventional period
* Self-reported history of hypertrophic obstructive cardiomyopathy, aortic valve stenosis, or mitral valve stenosis (since symptoms of these conditions may be aggravated by NTG therapy)
* Self-reported history of coronary disease (since patients with coronary disease may need NTG therapy for chest pain or may be at increased risk of new coronary events in the setting of nitrate tolerance), or evidence of prior myocardial infarction on screening electrocardiogram (ECG)
* Self-reported history of diabetes or 2 or more major risk factors for coronary disease (i.e., smoking, hypertension, or hyperlipidemia with physician-recommended pharmacologic treatment)
* Evidence of tachyarrhythmias such as atrial fibrillation or flutter without adequate rate control (>110 beats/minute) on screening ECG
* Evidence of second or third-degree atrioventricular block on screening ECG
* Hypotension based on measured resting blood pressure <90/60 at baseline; or normal resting blood pressure but evidence of orthostatic hypotension with change from supine to standing position)
* Uncontrolled hypertension based on measured resting blood pressure > 180/110 at baseline
* Self-reported headaches interfering with activities of daily activities more than twice a month, or use of prescription medication to prevent or treat headache in the past month (since these may be worsened by NTG therapy)
* Known allergy to nitroglycerin or other nitrate-based medications.
* Known skin sensitivity to adhesives (which may generalize to the NTG patches)
* Unable to complete or tolerate a brief 3-day run-in period involving the lowest available dose of NTG (0.1 mg/hr)
* Currently pregnant, gave birth within the past 3 months, planning pregnancy during the study period, or unwilling to use regular barrier contraception or abstain from sexual activity to prevent pregnancy if not yet postmenopausal
* Currently breastfeeding, breastfeeding within the past 3 months, or planning to breastfeed during the study period
* Self-report heavy alcohol use (>3 drinks in a given day or >7 drinks per week) and uncomfortable or unwilling to decrease their alcohol intake during the study period.
* Unable or unwilling to provide informed consent, fill out questionnaires, or complete study visits in English
* Report other conditions that, in the judgment of the investigators, render potential participants highly unlikely to follow the protocol, including plans to move, substance abuse, significant psychiatric problems, or severe dementia.

Ages: 40 Years to 62 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Huang, MD, MPhil, MAS, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, Oakland, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang AJ, Cummings SR, Ganz P, Schembri M, Raghunathan H, Vittinghoff E, Gibson CJ, Grady D. Efficacy of Continuous Transdermal Nitroglycerin for Treating Hot Flashes by Inducing Nitrate Cross-tolerance in Perimenopausal and Postmenopausal Women: A Randomized Clinical Trial. JAMA Intern Med. 2023 Aug 1;183(8):776-783. doi: 10.1001/jamainternmed.2023.1977. PMID 37273224

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transdermal Nitroglycerin | Placebo
Started | 70 | 71
Completed | 66 | 70
Not Completed | 4 | 1
Not completed — Cannot tolerate medication | 1 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Too busy | 1 | 0
Not completed — Incomplete outcome data | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transdermal Nitroglycerin | Placebo | Total
Number analyzed (Participants) | 70 | 71 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.27 (3.9) | 53.89 (3.8) | 54.57 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 71 | 141
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 4 | 16
  White | 50 | 50 | 100
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 70 | 71 | 141
Hot Flash Frequency (per day) [Mean (Standard Deviation); unit: episodes per day] | 10.77 (4.0) | 10.9 (2.9) | 10.84 (3.5)
Hot Flash Related Daily Interference Scale (HFRDIS) score [Mean (Standard Deviation); unit: units on a scale] — Range of 0-100. Higher score indicates lower quality of life.
  units on a scale | 46.11 (23.1) | 40.30 (21.0) | 43.18 (22.2)
Menopause Quality of Life (MENQOL), Vasomotor domain score [Mean (Standard Deviation); unit: units on a scale] — Range 1-8. Higher score indicates lower quality of life.
  units on a scale | 6.49 (23.1) | 6.21 (1.4) | 6.35 (1.4)
Pittsburgh Sleep Quality Index (PSQI) score [Mean (Standard Deviation); unit: units on a scale] — Range 0-21. Higher score indicates lower quality of life.
  units on a scale | 8.03 (3.7) | 7.74 (3.1) | 7.88 (3.4)
Generalized Anxiety Disorder-7 (GAD-7) score [Mean (Standard Deviation); unit: units on a scale] — Range 0-21. Higher score indicates lower quality of life.
  units on a scale | 3.13 (3.0) | 2.48 (3.0) | 2.80 (3.0)
Center for Epidemiologic Studies Depression (CES-D) Score [Mean (Standard Deviation); unit: units on a scale] — Range 0-60. Higher score indicates lower quality of life.
  units on a scale | 8.35 (6.8) | 8.9 (7.6) | 8.63 (7.1)
Moderate-to-severe hot flashes (per day) [Mean (Standard Deviation); unit: episodes per day] — Range 12-60, Higher score indicates lower quality of life.
  episodes per day | 8.68 (4.1) | 8.10 (3.0) | 8.39 (3.6)
Total hot flash severity score [Mean (Standard Deviation); unit: units on a scale] | 21.10 (9.1) | 20.42 (6.0) | 20.76 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Hot Flash Frequency
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 5 and 12 month time points.
Time Frame: Repeated change from baseline to 5 and 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Hot flashes per day
Arm/Group | Transdermal Nitroglycerin | Placebo
Number analyzed (Participants) | 66 | 70
Hot flashes per day | -4.56 [-6.01 to -3.11] | -4.02 [-5.41 to -2.63]
Statistical Analysis 1: Comparison: Transdermal Nitroglycerin vs Placebo; Test type: Superiority; p = 0.34, Mixed Models Analysis; Mixed Models adjusted for baseline value, age, race, and Hispanic ethnicity. Repeated measures mixed models, with unstructured co-variance matrix; Model generated Least Square Mean = -0.54, 95% CI 2-sided [-1.66 to 0.58] — Model generated LS Mean Differences

2. Secondary Outcome: Change From Baseline Hot Flash Related Daily Interference Scale (HFRDIS) Score
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 5 and 12 month time points.
  Range 0-100, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 5 and 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Transdermal Nitroglycerin | Placebo
Number analyzed (Participants) | 66 | 71
units on a scale | -19.85 [-28.5 to -11.2] | -20.36 [-28.61 to -12.12]
Statistical Analysis 1: Comparison: Transdermal Nitroglycerin vs Placebo; Test type: Superiority; p = 0.88, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Model generated Least Square Mean = 0.51, 95% CI 2-sided [-6.15 to 7.18] — Model generated LS Mean Differences

3. Secondary Outcome: Change From Baseline Menopause Quality of Life (MENQOL), Vasomotor Domain Score
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 5 and 12 month time points.
  Range 1-8, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 5 and 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Transdermal Nitroglycerin | Placebo
Number analyzed (Participants) | 66 | 71
units on a scale | -1.53 [-2.42 to -0.64] | -1.33 [-2.17 to -0.49]
Statistical Analysis 1: Comparison: Transdermal Nitroglycerin vs Placebo; Test type: Superiority; p = 0.57, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Model generated Least Square Mean = -0.2, 95% CI 2-sided [-0.88 to 0.48] — Model generated LS Mean Differences

4. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Score
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 5 and 12 month time points Range 0-21, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 5 and 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Transdermal Nitroglycerin | Placebo
Number analyzed (Participants) | 65 | 70
score on a scale | -1.27 [-2.23 to -0.31] | -1.18 [-2.1 to -0.26]
Statistical Analysis 1: Comparison: Transdermal Nitroglycerin vs Placebo; Test type: Superiority; p = 0.81, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Model generated Least Square Mean Differ = -0.09, 95% CI 2-sided [-0.8 to 0.63] — Model generated LS Mean Differences

5. Secondary Outcome: Change From Baseline Generalized Anxiety Disorder-7 (GAD-7) Score
Description: as for outcome 4
Time Frame: Repeated change from baseline to 5 and 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Transdermal Nitroglycerin | Placebo
Number analyzed (Participants) | 66 | 71
units on a scale | -0.15 [-1.18 to 0.89] | -0.57 [-1.56 to 0.42]
Statistical Analysis 1: Comparison: Transdermal Nitroglycerin vs Placebo; Test type: Superiority; p = 0.3, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Model generated Least Square Mean Differ = 0.43, 95% CI 2-sided [-0.38 to 1.23] — Model generated LS Mean Differences

6. Secondary Outcome: Change From Baseline Center for Epidemiologic Studies Depression (CES-D) Score
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 5 and 12 month time points Range 0-60, a higher score indicates a lower quality of life.
Time Frame: Repeated change from baseline to 5 and 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Transdermal Nitroglycerin | Placebo
Number analyzed (Participants) | 65 | 70
units on a scale | -1.39 [-3.89 to 1.11] | -1.79 [-4.18 to 0.6]
Statistical Analysis 1: Comparison: Transdermal Nitroglycerin vs Placebo; Test type: Superiority; p = 0.68, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Model generated Least Square Mean Differ = 0.4, 95% CI 2-sided [-1.52 to 2.32] — Model generated LS Mean Differences

7. Secondary Outcome: Change in Baseline Frequency of Moderate-to-severe Hot Flashes
Description: as for outcome 1
Time Frame: Repeated change from baseline to 5 and 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Hot flashes per day
Arm/Group | Transdermal Nitroglycerin | Placebo
Number analyzed (Participants) | 66 | 70
Hot flashes per day | -3.27 [-4.64 to -1.9] | -2.44 [-3.74 to -1.14]
Statistical Analysis 1: Comparison: Transdermal Nitroglycerin vs Placebo; Test type: Superiority; p = 0.12, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Model generated Least Square Mean Differ = -0.83, 95% CI 2-sided [-1.89 to 0.23] — Model generated LS Mean Differences

8. Secondary Outcome: Change in Baseline Total Hot Flash Severity Score
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 5 and 12 month time points. The hot flash severity score is calculated as the sum of severity ratings for all hot flashes recorded on the symptom over a 7-day period (mild=1, moderate=2, severe=3), and then divided by 7 for the daily average score.
  Range 12-60, higher score indicates lower quality of life.
Time Frame: Repeated change from baseline to 5 and 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Transdermal Nitroglycerin | Placebo
Number analyzed (Participants) | 66 | 70
units on a scale | -8.33 [-11.44 to -5.21] | -6.92 [-9.89 to -3.95]
Statistical Analysis 1: Comparison: Transdermal Nitroglycerin vs Placebo; Test type: Superiority; p = 0.25, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Model generated Least Square Mean Differ = -1.41, 95% CI 2-sided [-3.81 to 0.99] — Model generated LS Mean Differences

9. Other Pre Specified Outcome: Number of Participants With Treatment Related Severe Adverse Events Defined by Common Terminology Criteria for Adverse Events (CTCAE) Severity Grade 3 or Higher.
Description: Number of participants with treatment related severe adverse events defined by Common Terminology Criteria for Adverse Events (CTCAE) severity grade 3 or higher.
Time Frame: Baseline to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Transdermal Nitroglycerin | Placebo
Number analyzed (Participants) | 66 | 71
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Transdermal Nitroglycerin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/71
Other Adverse Events (participants affected / at risk) | 65/70 | 66/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Nitroglycerin (N=70) | Placebo (N=71)
Heart Fluttering (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (6) | 4 (5)
Soft Stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sore Tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach Discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upset Stomach (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Chest Pain Aggravated (General disorders) | 1 (1) | 0 (0)
Chest Pressure Sensation (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Feelings Of Weakness (General disorders) | 1 (1) | 0 (0)
Breast Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus Infection (Infections and infestations) | 0 (0) | 1 (1)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1)
Stomach Flu (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 7 (7) | 8 (9)
Accidental Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coccyx Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mosquito Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thigh Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arm Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back Ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hand Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid Arthritis Aggravated (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ductal Carcinoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (6) | 7 (9)
Headache (Nervous system disorders) | 58 (95) | 61 (101)
Lost Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Numbness Of Upper Extremities (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Taste Abnormality (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Depression Nos (Psychiatric disorders) | 1 (1) | 0 (0)
Emotional Distress (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Dyspareunia; Vaginal Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus Pressure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythematous Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Localised Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 17 (19)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Poison Oak Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritic Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Raynaud-Like Phenomena (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT02714205/Prot_SAP_000.pdf